CLINICAL TRIAL: NCT01978678
Title: Does Asthma Phenotype Have Impact on Disease Control - Can Detection of Inflammation and Hyper Responsiveness Ensure Stable Disease Faster
Brief Title: Does Asthma Phenotype Have Impact on Disease Control
Acronym: Aperitif
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Backer, DmSci, professor, md, Bispebjerg Hospital
Other Study IDs: Aperitif
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2013-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmicort: ICS and LABA - based on ACQ and FeNO
  Interventions: Drug: Pulmicort

INTERVENTIONS:
Drug: Pulmicort — ACQ and FeNO
  Other Names: RCT study

SUMMARY:
The application of biomarkers that are more closely associated with eosinophillic airway inflammation, such as measurements of FeNO level, cell count in induced sputum or bronchial reactivity could improve asthma control by better directing treatment. A systematic review and meta-analysis is to be conducted to assess the efficacy of tailoring asthma intervention on clinical symptoms compared with exhaled nitric oxide or induced sputum count.

DETAILED DESCRIPTION:
AHR used as outcome

ELIGIBILITY:
Inclusion Criteria:

* positiv mannitol
* asthma diagnose

Exclusion Criteria:

* other lung disease

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly referred asthma patients
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Control of asthma based on an algorithm | 2 years
  Based on ACQ and FeNO

SECONDARY OUTCOMES:
The use of NO and sputum cell count as a marker in asthma management | 2 years
  Based on ACQ and FeNO

OTHER OUTCOMES:
the use of ACQ and miniAQLQ | 2 years
  Based on ACQ and FeNO

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, MD, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Department of Respiratory Medicine, L, Bispebjerg Hospital,, Copenhagen, NV
  - Respiratory research unit, Bispebjerg University Hospital, Copenhagen